CLINICAL TRIAL: NCT05416554
Title: Long-term Cognitive, Neuropsychiatric and Functional Outcomes in Adults Who Have Received Chimeric Antigen-Receptor T-Cell (CAR-T) Therapy for Aggressive Lymphoma at Stanford - A Pilot Study
Brief Title: Long-term Cognitive, Neuropsychiatric and Functional Outcomes in Adults Who Have Received Chimeric Antigen-Receptor T-Cell (CAR-T) Therapy for Aggressive Lymphoma at Stanford
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-56813; CCT5069 (Other: OnCore)
Record Dates: First submitted 2022-05-20; First posted 2022-06-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuropsychological testing (Other): Participants will take neuropsychological testing in-person or via telehealth video
  Interventions: Behavioral: Neuropsychological testing

INTERVENTIONS:
Behavioral: Neuropsychological testing — Upon completion of the consent, the subject will be booked into an available 90 minute in-person or remote neuropsychological testing

SUMMARY:
This study aims to assess the feasibility of performing neuropsychological testing to measure the cognitive performance of individuals following Axicabtagene ciloleucel CAR-T therapy at Stanford.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years-old
* Treated with Axicabtagene ciloleucel CAR-T therapy at Stanford Or
* Treated with standard commercial Axicabtagene ciloleucel CAR-T therapy elsewhere and followed primarily by SHC Blood and Bone Marrow transplant providers
* >/= 6 months from the date of CAR-T infusion
* Fluent in English
* Able to attend and participate in in-person testing (Arm I)
* Able to participate in remote video testing with adequate workspace, computer and internet capabilities for a reliable telehealth video connection (Arm II)

Exclusion Criteria:

* Concurrent enrollment in a CAR-T therapeutics research study
* Unable to be present for the scheduled testing
* Unable to participate in testing due to severe cognitive or physical limitation
* Actively receiving chemotherapy
* Progressive cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who complete neuropsychological testing in the post-CAR-T adult population | 6 months
Number of patients who complete telehealth neuropsychological testing in the post-CAR-T adult | 6 months

SECONDARY OUTCOMES:
Wechsler Test of Adult Reading WTAR Neuropsychological testing | Baseline
  The neuropsychological testing will capture any potential deficits in language, processing speed, executive functioning and visuospatial abilities, and may be compared to age and education-matched normative data.
Hopkins Verbal Learning Test HVLT | Baseline
  The neuropsychological testing will capture any potential deficits in language, processing speed, executive functioning and visuospatial abilities, and may be compared to age and education-matched normative data.
Controlled Oral Work Association Test COWAT | Baseline
  The neuropsychological testing will capture any potential deficits in language, processing speed, executive functioning and visuospatial abilities, and may be compared to age and education-matched normative data.
Trails A and B (Oral Trails) | Baseline
  The neuropsychological testing will capture any potential deficits in language, processing speed, executive functioning and visuospatial abilities, and may be compared to age and education-matched normative data.
Digit Span | Baseline
  The neuropsychological testing will capture any potential deficits in language, processing speed, executive functioning and visuospatial abilities, and may be compared to age and education-matched normative data.
Clock Drawing Test | Baseline
  The neuropsychological testing will capture any potential deficits in language, processing speed, executive functioning and visuospatial abilities, and may be compared to age and education-matched normative data.
Short form of Quality of Life SF-36 | Baseline
  Items from the SF36 (Short Form 36) survey
General Anxiety Disorder Assessment GAD-7 | Baseline
  Assesses anxiety symptoms
  The following cut-offs correlate with level of anxiety severity:
  Score 0-4: Minimal Anxiety, Score 5-9: Mild Anxiety, Score 10-14: Moderate Anxiety, Score greater than 15: Severe Anxiety
Patient Health Questionnaire PHQ9 | Baseline
  Assesses depressive symptoms PHQ-9 Score 0 - 4 None, Mild= 5 - 9 , Moderate=10 - 14 , Moderately Severe=15 - 19 , Severe=20 - 27

CONTACTS AND LOCATIONS:
Overall Officials: Brian Scott, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, San Francisco, California, United States